CLINICAL TRIAL: NCT03025009
Title: A Single-Site, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Glucodynamic Effects of LY3192767 in Healthy Subjects
Brief Title: A Study of LY3192767 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16242; I8M-MC-BIXA (Other: Eli Lilly and Company); 2016-003274-40 (EudraCT Number)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — basal insulin peglispro; LY2605541; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY3192767 (Part A) (Experimental): Escalating doses of LY3192767 administered subcutaneously (SC).
  Interventions: Drug: LY3192767
- Placebo (Part A) (Placebo Comparator): Placebo matching LY3192767 administered subcutaneously (SC).
  Interventions: Drug: Placebo
- LY3192767 (Part B) (Experimental): LY3192767 administered as a SC injection in one of three study periods.
  Interventions: Drug: LY3192767
- Basal Insulin Peglispro (Part B) (Active Comparator): Basal insulin peglispro administered as a SC injection in one of three study periods.
  Interventions: Drug: Basal Insulin Peglispro
- Insulin Glargine (Part B) (Active Comparator): Insulin glargine administered as a SC injection in one of three study periods.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY3192767 — Administered SC.
  Arms: LY3192767 (Part A); LY3192767 (Part B)
Drug: Basal Insulin Peglispro — Administered SC.
  Other Names: LY2605541
  Arms: Basal Insulin Peglispro (Part B)
Drug: Insulin Glargine — Administered SC.
  Arms: Insulin Glargine (Part B)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A)

SUMMARY:
The main purpose of this study is to investigate the side effects related to LY3192767 when given as an injection under the skin to healthy participants. Blood tests will be done to check how much LY3192767 is absorbed into the bloodstream, how long it takes for the body to get rid of it, and how it affects blood sugar levels. The study has two parts: Part A and Part B. Each participant will enroll in one part. For each participant, Part A will last up to about 32 days after last dose and Part B will last up to about 49 days after last dose. Screening must be completed prior to study start.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Have a body mass index (BMI) of >18.5 and <30.0 kilogram per square meter (kg/m²), inclusive

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have participated as a participant in a first-in-human study within 90 days of the initial dose of study drug
* Have known allergies to insulin, heparin, or related drugs, or history of relevant allergic reactions of any origin
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, chronic inflammatory disease, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Study Completion (up to about Day 49)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of LY3192767 | Predose through 336 Hours
  PK: Tmax of LY3192767
PK: Maximum Serum Concentration (Cmax) of LY3192767 | Predose through 336 Hours
  PK: Cmax of LY3192767
PK: Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC[0-inf] of LY3192767 | Predose through 336 Hours
  PK: AUC(0-inf) of LY3192767
Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot) of LY3192767 | Predose through 36 Hours During Clamp Procedure
  PD: Total Amount of Glucose Infused (Gtot) of LY3192767
PD: Maximum Glucose Infusion Rate (Rmax) of LY3192767 | Predose through 36 Hours During Clamp Procedure
  PD: Rmax of LY3192767
PD: Time of Maximum Glucose Infusion Rate (TRmax) of LY3192767 | Predose through 36 Hours During Clamp Procedure
  PD: TRmax of LY3192767
PD: Change from Baseline in Free Fatty Acids | Predose through 48 Hours Postdose
  PD: Change from Baseline in Free Fatty Acids
PD: Change from Baseline in Glycerol | Predose through 48 Hours Postdose
  PD: Change from Baseline in Glycerol
PD: Change from Baseline in Triglycerides | Predose through 48 Hours Postdose
  PD: Change from Baseline in Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No